CLINICAL TRIAL: NCT01993784
Title: Phase IIa Study of Nimotuzumab in Second or Late- Line Treatment of Patients With Locally Advanced or Metastatic Esophageal Squamous Cell Carcinomas
Brief Title: Study of Nimotuzumab to Treat Esophageal Squamous Cell Carcinoma.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, Department of GI Oncology,Peking University, School of Oncology, Beijing Cancer Hospital & Institute, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESCC-N-301
Record Dates: First submitted 2013-08-16; First posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Esophageal Squamous Cell Cancer
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — nimotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nimotuzumab (Experimental): the nimotuzumab treatment: 2 levels (400 mg/w, 600 mg/w, weekly, until disease progression)
  Interventions: Drug: nimotuzumab

INTERVENTIONS:
Drug: nimotuzumab

SUMMARY:
Nimotuzumab is an IgG1 humanized monoclonal antibody that recognized an epitope located in the extra cellular domain of the human epidermal growth factor receptor (EGFR). Clinical efficacy has been shown in adult with head and neck cancer. The study assessed the safety and efficacy of different dosage of Nimotuzumab in second or late- line treatment of patients with locally advanced or metastatic esophageal squamous cell carcinomas.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed esophageal squamous carcinoma,failed to first or second line chemothrepay
* Age 18 to 75 years old
* Measurable disease according to the RECIST criteria(diameter of the lesion should be more than 10mm by spiral CT or MRI, more than 20mm by common CT, the date of image should be less than 15 days before enrollment)
* Life expectancy of ≥3 month
* Karnofsky performance status ≥80
* WBC>3,000/mm3, absolute neutrophil count ≥1500/mm3, platelet>100,000/mm3, Hb>9g/dl，Bilirubin level < 1.0 times ULN，Serum creatinine <1.0 times ULN，ALT and AST<2.5 times ULN ，AKP < 2.5 times ULN ，(≤5 times ULN in patients with liver metastases)(within 7 days before enrollment)
* No sever complication, such as active gastrointestinal bleeding, perforation, jaundice, obstruction, non-cancerous fever>38℃；
* Normal ECG/cardiac function
* Good compliance
* Having signed informed consent -

Exclusion Criteria:

* No previous systemic therapy for metastatic esophageal squamous carcinoma
* Known hypersensitivity to study drugs
* Tumor with length≥10cm, liver metastasis covers more than 50% of liver,or lung metastasis covers more than 25% of lung
* No measurable lesions, eg. pleural fluid and ascites
* Only with Other previous malignancy within 5 year, except non-melanoma skin cancer
* Heart failure or other sever organ dysfunction, eg. coronary artery disease, myocardial infarction within the last 6 months only Brain or bone metastasis
* Chronic diarrhea
* Mentally abnormal or disable cognition,including CNS metastasis
* Pregnancy or lactation period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-03 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 6 weeks
  CT/MRI will be performed every 2 cycles of treatment for efficacy evaluation

SECONDARY OUTCOMES:
adverse events | during the treatment in the hosptital,an expected average of 1 week
  participants will be followed for the duration of hospital stay, an expected average of 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, MD, Principal Investigator — Peking Universtiy Cancer Hospital
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China